CLINICAL TRIAL: NCT00757874
Title: A Double Blind Phase II Study Comparing Safety and Efficacy of Tacrolimus Versus Topical Clobetasol Propionate in the Treatment of Vulvar Lichen Sclerosus.
Brief Title: Tacrolimus Versus Clobetasol Propionate in the Treatment of Vulvar Lichen Sclerosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deana Funaro (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Deana Funaro, Dermatologist, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StJustineH
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Female urogenital disease; skin disease
MeSH Terms: conditions — Vulvar Lichen Sclerosus; Female Urogenital Diseases; Skin Diseases | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus cream (Experimental)
  Interventions: Drug: Tacrolimus cream
- Clobetasol cream (Active Comparator)
  Interventions: Drug: Clobetasol cream

INTERVENTIONS:
Drug: Tacrolimus cream — 0.5 g per day at bed time for 3 months or less.
  Other Names: Prtopic
  Arms: Tacrolimus cream
Drug: Clobetasol cream — 0.5 gram each day at bed time during 3 months or less.
  Other Names: Dermovate
  Arms: Clobetasol cream

SUMMARY:
Lichen Sclerosus is an inflammatory skin condition affecting mostly the genital area of persons of all ages, gender or race. The most frequent complaint is that of itchiness of the vulva but pain may also occur. Some women will experience no symptoms at all. However, it is important to treat this condition since it may increase and cause important scarring and deformity. In less than 5% of cases, cancer may develop.

Lichen Sclerosus is a chronic disease which can be controlled but not cured. Topical corticosteroids are the usual treatment for this condition. Though this treatment is generally well tolerated, some patients may not present a sufficient response or may develop mainly local and rarely systemic side effects. In this perspective, an alternative treatment would be beneficial.

Tacrolimus, a topical immunomodulator has been approved for the treatment of atopic eczema and has shown its efficacy in the treatment of vulvar lichen sclerosus in a limited number of patients. Tacrolimus acts as a non-steroidal anti-inflammatory agent (NSAI) without causing the usual side effects seen with the prolonged use of topical corticosteroids.

This study is designed to evaluate the safety and efficacy of tacrolimus in treating vulvar lichen sclerosus by comparing it with the standard topical corticosteroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female, 2 years or older
* Medical diagnosis of vulvar lichen sclerosus
* Received no treatment during the last 4 weeks

Exclusion Criteria:

* Who have received topical steroids, tacrolimus or pimecrolimus during the 4 last weeks.
* Who are immunocompromised
* Who have history of intra-epithelial neoplasia or anogenital carcinoma
* Who have active vulvar infections (herpes,condylomas,vaginitis)
* Who are hypersensitive to tacrolimus, pimecrolimus or corticosteroids
* Who have physical limitations that cause difficulty in applying the cream
* Who wear diapers
* Who present Hyperkeratotic Vulvar Lichen Sclerosus

Min Age: 2 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-04; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To document the efficacy of Tacrolimus vs topical clobetasol propionate in the treatment of Vulvar Lichen Sclerosus by medical examinations and reporting of the symptoms. Cream is applied once a day for 3 months | Comparison before the treatment and monthly for 3 months.

SECONDARY OUTCOMES:
Compared presence and severity of side effects of both groups. | During the 3 months of treatment
CBC, Glycemia, vitamine B 12 dosage, TSH (to find associated auto-immune diseases) | At 1 to 3 months after starting the study, collected once.

CONTACTS AND LOCATIONS:
Overall Officials: Deana Funaro, Doctor, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada